CLINICAL TRIAL: NCT06467539
Title: Novel Augmentation of DAOIB and Antioxidant for Early Dementia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 202200458A3C502
Record Dates: First submitted 2024-06-16; First posted 2024-06-21 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Mild Cognitive Impairment
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): DAOIB plus Antioxidant agent (AO)
  Interventions: Drug: DAOIB plus AO
- Placebo Comparator (Placebo Comparator): DAOIB plus Placebo
  Interventions: Drug: DAOIB plus placebo

INTERVENTIONS:
Drug: DAOIB plus AO — oral, for 24 weeks
  Arms: Experimental
Drug: DAOIB plus placebo — oral, for 24 weeks
  Arms: Placebo Comparator

SUMMARY:
Previous studies found that some NMDA-enhancing agents were able to improve cognitive function of patients with early-phase dementia. In addition, several drugs with antioxidant properties have been tested in clinical trials for the treatment of dementia too. Whether combined treatment of an NMDA-enhancing agent and a drug with antioxidant property can be better than an NMDA-enhancing agent alone deserves study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's disease or mild cognitive impairment
* MMSE between 10-26
* CDR 1 or 0.5

Exclusion Criteria:

* Hachinski Ischemic Score > 4
* Substance abuse/dependence
* Parkinson disease, epilepsy, dementia with psychotic features
* Major depressive disorder
* Major physical illnesses
* Severe visual or hearing impairment

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the Alzheimer's disease assessment scale - cognitive subscale at week 8, 16 and 24 | week 0, 8, 16, 24
  Alzheimer's disease assessment scale-cognitive subscale consists of 11 tasks. Its scores range from 0 (best) to 70 (worst).

SECONDARY OUTCOMES:
Change from baseline in Clinician's Interview-Based Impression of Change plus Caregiver Input score at week 8, 16 and 24 | week 8, 16, 24
  Clinician's Interview-Based Impression of Change plus Caregiver Input score is a global assessment of change based on a comprehensive, semi-structured interview which includes caregiver-supplied information. It is a 7-point rating scale ranging from 1-7, where 1 represents markedly improved; 4, no change; and 7, markedly worse.
Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24 | week 0, 8, 16, 24
  Change from baseline in Mini-Mental Status examination score at week 8, 16 and 24
Change from baseline in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) score at week 8, 16 and 24 | week 0, 8, 16, 24
  Clinical Dementia Rating Scale (CDR) is a global assessment tool that yields global and Sum of Boxes scores (SB). Compared to the global CDR score, the CDR-SB score provides better utility in tracking changes in dementia severity.
Change from baseline in Alzheimer's disease Cooperative Study scale for ADL in MCI (ADCS-MCI-ADL) score at week 8, 16 and 24 | week 0, 8, 16, 24
  ADCS-MCI-ADL appears to be a suitable instrument for evaluating activities of daily living in mild cognitive impairment. Its scores range from 0 (worst) to 78 (best).
Change from baseline in Medical Outcomes Study Short-Form-36 (SF-36) score at week 8, 16 and 24 | week 0, 8, 16, 24
  The SF-36 consists of eight sections which assess the quality of life.
Change from baseline in the composite score of a battery of additional cognitive tests at week 8, 16 and 24 | week 0, 24
  The battery of additional cognitive tests include speed of processing (Category Fluency), working memory (verbal and nonverbal, Wechsler Memory Scale), learning and memory tests (verbal and visual, Wechsler Memory Scale).

CONTACTS AND LOCATIONS:
Locations (1):
- Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No